CLINICAL TRIAL: NCT03288909
Title: Ultra High Field Magnetic Resonance Imaging as a Biomarker for Premotor Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Matthew Brodsky, Associate Professor of Neurology, Oregon Health and Science University
Other Study IDs: eIRB#5611
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Parkinson Disease; REM Sleep Behavior Disorder
MeSH Terms: conditions — Parkinson Disease; REM Sleep Behavior Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Early onset Parkinson's disease: Idiopathic Parkinson's disease within 1 year of symptom onset
  Interventions: Other: MRI
- Idiopathic REM Sleep Behavior Disorder: Idiopathic REM Sleep Behavior Disorder
  Interventions: Other: MRI
- Age-matched healthy controls: Age-matched healthy controls
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI

SUMMARY:
This is a prospective observational study investigating the utility of 7 Tesla MRI to quantify nigrosome1 signal in a cohort of individuals with recent onset Parkinson's disease and in at-risk cohorts at a premotor state of Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease within 1 year of motor symptom onset. Idiopathic REM sleep behavior disorder without signs/symptoms of Parkinson's disease.

Age-matched controls.

Exclusion Criteria:

* Atypical Parkinsonism
* Contraindications for MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Idiopathic Parkinson's disease within 1 year of motor symptom onset. Idiopathic REM sleep behavior disorder without signs/symptoms of Parkinson's disease.
  Age-matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2015-09; Primary Completion 2020-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative signal analysis of nigrosome 1 | 1 year

SECONDARY OUTCOMES:
Change in quantitative signal analysis of nigrosome 1 | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Brodsky, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided